CLINICAL TRIAL: NCT06181929
Title: A Prospective Study for the Early Diagnosis of Lung Cancer in Korean Females Who Are Never Smoker with a Family History of Lung Cancer
Brief Title: A Prospective Study for the Early Diagnosis of Lung Cancer in Korean Females
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Sang-Won Um (Other)
Responsible Party: Sponsor-Investigator, Sang-Won Um, professor, Samsung Medical Center
Organization: Samsung Medical Center (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 20223-10-101
Record Dates: First submitted 2023-11-09; First posted 2023-12-26 (Actual); Last update posted 2025-03-05 (Actual); Status verified 2024-03

CONDITIONS: Health Risk Behaviors
MeSH Terms: conditions — Health Risk Behaviors

STUDY DESIGN:
Intervention Model Description: single-arm prospective pilot study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- intervation group (Experimental): LDCT screening exam
  Interventions: Diagnostic Test: Low dose CT

INTERVENTIONS:
Diagnostic Test: Low dose CT — A subject can voluntarily discontinue active screening with LDCTs after the baseline LDCT is completed but will remain in study follow-up with follow-up calls in 12-month intervals for up to 10 years since initial consent

SUMMARY:
This is a single-arm prospective pilot study in a single institution. The target accrual is 200 participants of Korean, female sex, never smoker status, and family history of lung cancer. The study will aim to enroll 200 participants in two years.

DETAILED DESCRIPTION:
Interested individuals will contact a research coordinator who will help to assess for study eligibility. Individuals who are eligible and able to sign informed consent will then proceed to have a LDCT screening exam with a result reported by a radiologist approved to read lung cancer screening scans. Results of this screening test will be discussed with the subject and further recommendations will be given. Negative results will proceed to have repeat LDCT exams for two additional years. Positive results will be recommended to have further diagnostic work-up, and possible treatment. Those with positive findings may be recommended to repeat a LDCT at varied intervals (e.g. at 3 months, at 6 months, etc.) per Lung-RADS recommendations which can be conducted as a research LDCT or as standard-of-care.

In addition, blood draw collection for a plasma-based assay will be collected at baseline, first year and second year for all patients along with the repeated LDCT scans.

A medical history questionnaire containing questions regarding ethnicity, family history of lung cancer, environmental exposures including secondhand smoke exposure, and a residential district to estimate the exposure of PM2.5 or PM10 will be given to the patient at the initial visit after informed consent has been obtained (Appendix A). Questionnaire can be collected within 1 month from the baseline consent.

ELIGIBILITY:
Inclusion Criteria:

1. Age 45-74 years old
2. Korean female
3. Never smoker defined as a lifetime exposure of less than 100 cigarettes
4. Family history of lung cancer at first degree relatives (parents, siblings, or children)

Exclusion Criteria:

1. Prior history of lung cancer.
2. Diagnosis of any cancer within the past five years
3. Participation in a cancer prevention trial.
4. Present symptoms suggestive of current lung cancer, including: unexplained weight loss of over 5 kilograms within the last 12 months or unexplained hemoptysis.
5. Medical or psychiatric condition precluding informed medical consent.
6. History of LDCT screening, chest CT, PET or PET/CT scan within 10 years

Ages: 45 Years to 74 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Korean female
Enrollment: 200 (Estimated)
Dates: Start 2024-06-01 (Actual); Primary Completion 2026-05-31 (Estimated); Study Completion 2034-05-31 (Estimated)

PRIMARY OUTCOMES:
Lung cancer detection rate | up to 2years
  detection rate

SECONDARY OUTCOMES:
incidence of lung cancer | up to 2years
  Whether lung cancer is found in each screening test conducted for the first (baseline) and first and second years
distribution of lung cancer stages | up to 2years
  number of lung cancer diagnosed, number of stage I, rate of surgery, rate of false positive
Estimation of the Early Detection Rate of Lung Cancer in Liquid Biopsy | up to 2years
  cfDNA

OTHER OUTCOMES:
identification of potential predictive biomarkers of malignancy | up to 2years
  EGFR mutation

CONTACTS AND LOCATIONS:
Overall Officials: Um Sang-Won, PhD, Principal Investigator — Samsung Medical Center
Locations (1):
- Samsung Medical Center, Seoul, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No